CLINICAL TRIAL: NCT05219097
Title: Comparison of the Specificity, Sensitivity and Clinical Correlation of CBA, RIPA and ELISA Assay in Detecting AChR and MuSK IgG of Myasthenia Gravis: a National Multicenter Study
Brief Title: The Specificity, Sensitivity and Clinical Correlation of CBA, RIPA and ELISA in Detecting AChR and MuSK IgG of Myasthenia Gravis
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Fu-Dong Shi, Professor, Tianjin Medical University General Hospital
Other Study IDs: IRB2021-YX-260-01
Record Dates: First submitted 2022-01-20; First posted 2022-02-01 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Detection Autoantibody of Myasthenia Gravis
Keywords: Cell-based assay; Radioimmunoprecipitation assay (RIPA); Enzyme-linked immunosorbent assay (ELISA); Autoantibody determination; Myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — sreum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cell Based Assay (CBA): Use AChR/MuSK Ab CBA Kit (Tianjin New Terrain Biological Technology Co., Ltd, China) to detect AChR and MuSK Ab of myasthenia gravis
  Interventions: Diagnostic Test: CBA Assay
- RIPA Assay: Use AChR and MuSK Ab radioimmunoassay kit (RSR Limited, UK) to detect AChR and MuSK Ab of myasthenia gravis
  Interventions: Diagnostic Test: CBA Assay
- ELISA Assay: Use AChR Ab ELISA Kit (RSR Limited, UK) and MuSK ELISA kit (IBL Limited, Germany) to detect AChR and MuSK Ab of myasthenia gravis
  Interventions: Diagnostic Test: CBA Assay

INTERVENTIONS:
Diagnostic Test: CBA Assay — Comparsion of specificity, sensitivity and clinical correlation of CBA, ELISA and RIPA assay in autoantibodies detection of myasthenia gravis
  Other Names: ELISA Assay; RIPA Assay

SUMMARY:
Myasthenia gravis (MG) is a neuromuscular junction (NMJ) disorder mediated by autoantibodies against AChR, MuSK or other autoantigens located at the post synaptic membrane of the neuromuscular junction. Presence of autoantibodies specific for AChR or MuSK can establish diagnosis in conjunction with clinical presentations. In most established guidelines for the diagnosis and treatment of myasthenia gravis, determination of AChR and MuSK antibodies has been recommended. Radioimmunoprecipitation assay (RIPA), enzyme-linked immunosorbent assay (ELISA), and cell-based assay (CBA) are all commercially available and have been adopted for autoantibody detection by most referring neurologists. At present, specificity and sensitivity of these methods have not been compared in large cohorts within a context of stringent quality control. As a consequence, there are no national or international consensus regarding selection of methods and interpretation of results, resulting in challenges to neurologists managing these patients. To this end, the investigators proposed to conduct a multicenter, double-blind, prospective study to compare the sensitivity and specificity of CBA, RIPA and ELISA assays to detect AChR and MuSK antibodies.

DETAILED DESCRIPTION:
Participants: patients with suspected MG

Aim: the specificity, sensitivity, and clinical correlation of AChR and MuSK IgG detection through the CBA, ELISA, and RIPA methods.

Study design: A multicenter, double-blind, prospective study to compare the sensitivity and specificity of CBA, RIPA, and ELISA assays in detecting AChR and MuSK antibodies.

Total enrollment: 3000 patients with suspected MG will be enrolled.

Time frame: The enrollment time of this trial is 21 months, and the entire study period is about 24 months.

Reagent resource: 1. Acetylcholine receptor autoantibody RIA kit: RSR limited, recommended cut-off value=0.5 nmol/L.

2. Acetylcholine receptor autoantibody CBA kit: Tianjin New Terrain Biological Technology Co., Ltd; recommended cut-off value =1:10.

3. Acetylcholine receptor autoantibody ELISA kit: RSR limited; recommended cut-off value=0.45 nmol/L.

4. Muscle-specific tyrosine kinase RIA kit: RSR limited, recommended cut-off value =0.05 nmol/L.

5. Muscle-specific tyrosine kinase CBA kit: Tianjin New Terrain Biological Technology Co., Ltd; recommended cut-off value =1:10.

6. Muscle-specific tyrosine kinase ELISA kit: IBL, recommended cut-off value=0.4 U/ml.

Groups: The samples were divided into 3 groups according to the detected methods: CBA group, RIPA group and ELISA group.

Study protocol: 1. When patients suspected of MG matched up with the inclusion and exclusion criteria, the serum sample of each patient would be divided into equal aliquots and randomly assigned to the CBA, ELISA, and RIPA testing laboratories for detection.

2. All patient's information will be masked and monitored by members of ethics committees. Serum specimens from participants will be renumbered without any clinical information before doing the tests to be investigated. According to the standard procedure of kits, the operator in laboratories to perform the CBA, ELISA, or RIPA will complete the detection of AChR and MuSK antibodies of the enrolled participants' serum, and record the original value, control, or reference value.

3. Each MG center will provide the clinical diagnosis results of the enrolled patients, treatment and follow up information of the participants. The diagnosis of MG and the tests to be investigated will be double blindly done.

4. The data statistics, analysis, and summary of the project are operated by an independent third-party statistic team.

Evaluation indicators: Evaluate the specificity, sensitivity, and clinical correlation of AChR and MuSK IgG detection through the CBA, ELISA, and RIPA methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with compatible clinical features of weakness of skeletal muscles, including ptosis, diplopia, dysphonia, dysphagia, or limb weakness.
* Patients need to do the diagnosis of MG, requiring serum autoantibody, electrophysiological, pharmacological neostigmine test, thymic computed tomography (CT) and magnetic resonance imaging (MRI), etc in the diagnostic evaluation of MG.

Exclusion Criteria:

* Patients with uncertain diagnoses or incomplete clinical data for data analysis.
* Patients with abnormal serum samples, such as hemolysis or lipemia, which will affect the detection base value and the final interpretation of CBA, RIPA and ELISA.

Ages: 1 Year to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected MG, 1-90 years of age.
Sampling Method: Probability Sample
Enrollment: 2663 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Comparsion of the specificity, sensitivity and clinical correlation | 24 months
  Comparsion the specificity,sensitivity and clinical correlation of CBA, RIPA and ELISA assay in autoantibodies detection of myasthenia gravis

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Dong Shi, MD, Ph.D, Study Chair — Beijing Tiantan Hospital,Tianjin Medical University General Hospital
Locations (2):
- China (2):
  - Beijing Tiantan Hospital, Beijing
  - Tianjin Medical University General Hospital, Tianjin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Z, Zhang C, Chang T, Zhang X, Yang H, Gao F, Feng J, Liu H, Chen S, Wang L, Yang C, Li H, Pan Y, Palace J, Shi FD; SCREAM Study Investigators. A multicentre, prospective, double-blind study comparing the accuracy of autoantibody diagnostic assays in myasthenia gravis: the SCREAM study. Lancet Reg Health West Pac. 2023 Jul 19;38:100846. doi: 10.1016/j.lanwpc.2023.100846. eCollection 2023 Sep. PMID 37554174